CLINICAL TRIAL: NCT06261697
Title: A Web-based Survey -Relationship Between Smartphone Addiction and Temporomandibular Joint Disorders Among Adults in Egypt: Cross Sectional Study
Brief Title: Relationship Between Smartphone Addiction and Temporomandibular Joint Disorders Among Adults in Egypt.
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Norhan Mohamed Eltayeb, principal investigator, Cairo University
Other Study IDs: P.T.REC/012/004876
Record Dates: First submitted 2024-01-25; First posted 2024-02-15 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Temporomandibular Disorders; Smartphone Addiction
Keywords: TMJ disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders; Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: A web based survey — An online based questionnaire includes three screens, the first includes the consent form, the second includes the demographic data , and the third page includes questionnaires
  Other Names: An online based questionnaire

SUMMARY:
Cross sectional study to investigate the relation between Smartphone addiction and temporomandibular disorders among youth population in Egypt. An online- based questionnaire study. A 296 participants who are Egyptians with age between18 and 35 years old without prior neck and upper extremity related diseases, orofacial trauma or surgeries, history of rheumatoid arthritis or congenital musculoskeletal problems. An online- based questionnaire will be sent through different social media platforms, it will include three screens, the first includes the consent form, the second includes the demographic data (year of birth, current educational status, gender and geographic information ), and the third page includes questionnaires

.

ELIGIBILITY:
Inclusion Criteria:

* both males and females adults
* Their ages between18 and 35 years old
* ability to use Smartphone

Exclusion Criteria:

* any neck and upper extremity related diseases
* orofacial trauma or surgeries
* history of Rheumatoid arthritis
* congenital musculoskeletal problems.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 296 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Fonseca Anamnestic Index (FAI) questionnaire | 2 months
  a questionnaire used to assess the severity of TMD
Smartphone Addiction Scale-Short version (SAS-SV) questionnaire | 2 months
  a questionnaire used to measure the degree of smartphone addiction
Patient Health Questionnaire (PHQ) | 2 months
  a questionnaire used to indicate the severity of depression